Abbreviated Title: Improving Patient Experience:

**BMBA** 

40

41

**Purpose** 

Version Number: 1.1 

Version Date: 01/10/2022

#### Jefferson Office of Human Research 1 2 **Informed Consent OHR-8** 3 Version Date – FOR OHR USE: 5/22/20 4 5 **Department**: Oncology Nursing 6 7 Principal Investigator: Anne Delengowski, RN, MSN, AOCN, CCCTM 8 9 Study Title: Improving the Patient Experience During Bone Marrow Biopsy/Aspiration (BMBA): 10 Do Interventions Decrease Distress and Pain. 11 12 Lay Title: Improving Patient Experience During Bone Marrow Biopsies 13 14 **General Information Section** 15 16 **Informed Consent** 17 18 You are being asked to take part in a research study. Research is different from standard 19 medical care, and is done to learn something new. 20 21 Please read on to find out: 22 23 • The purpose of this research. 24 How this research is different from standard medical care. 25 • The procedures involved. 26 • The risks. 27 • The possible benefits. 28 The alternatives to taking part in this research. 29 30 You will have the opportunity to discuss this study with the research personnel. Use this 31 information to decide if you want to take part in this research. This process is called informed 32 consent. 33 34 **Voluntary Participation** 35 36 You do not have to take part in this research. It is your choice whether or not you want to take 37 part. If you choose not to take part or choose to stop taking part at any time, there will be no 38 penalty or loss of benefits that you would normally get. 39

Approved until END OF STUDY

APPROVAL DATE 10/28/2021

THOMAS JEFFERSON UNIVERSITY IRB

PI: Anne Delengowski, RN, MSN, AOCN, CCCTM

IRB Control #: 21G.1035

Abbreviated Title: Improving Patient Experience:

BMBA

Version Number: 1.1 

Version Date: 01/10/2022

The purpose of this research is to explore ways of improving the patient experience during visits for bone marrow biopsies. This procedure can be painful and cause distress. This study will look at alternative ways of promoting relaxation and distraction both while waiting before the

procedure and during the procedure.

45 46 47

## How this Research is Different from Standard Medical Care

48 49

50

51

52

Depending on which group you are assigned to, you may receive different tools to help promote relaxation and reduce distress during your procedure. These include changes to the room environment, music, guided meditation, and virtual reality. These are all techniques that have been used to help reduce pain and distress for cancer patients, but they have not been specifically used during bone marrow biopsies.

535455

## **Number of Participants**

5657

About 60 people will take part in this research in the whole study at Jefferson.

58 59

#### **Duration**

60 61

You will be in this research study for a single bone marrow biopsy procedure visit.

62 63

# **Procedures and Risks**

64 65

It is important that you know the procedures and risks involved in this research. These will be discussed with you and are included in detail later in this form. Review the information carefully when making your decision to take part in this research.

67 68 69

66

## **Possible Benefits**

70 71

72

73

You may personally benefit from taking part in this research. Some of the possible benefits may be decreased distress, decreased pain, and improved satisfaction. Your participation will help us understand what methods are best to improve the overall patient experience during this procedure.

747576

# **Alternatives to Taking Part in this Research**

77 78

The alternative to being in this study is to not take part.

79 80

# **Payment**

Abbreviated Title: Improving Patient Experience:

**BMBA** 

You will not be paid for taking part in this study. If this research or the information or specimens you provide result in commercial profit, you will not receive any money from that profit.

Version Date: 01/10/2022

Version Number: 1.1


# **Ending Study Early**

There are a number of reasons you may decide or be asked to stop the study early (example: medical issues). You may also have to stop the study early even if you do not want to. You and the research personnel will discuss the reason if this becomes necessary. If you do leave the study early, you may be asked to complete some of the procedures described in this form. This will include completing the post-procedure survey.

#### **New Information**

New information may come out during this study. You will be given any new information that could change your decision to take part. You may ask to see the information collected about you, but not until the entire study is complete. You will be given any research results that could affect your health.

# **Detailed Information Section**

## **Drugs/Devices**

The two interventions used in this study are described below:

Intervention 1 uses a virtual reality headset to provide a guided meditation experience. Virtual reality, or VR, is a simulated experience that combines going to a movie with the interactions of playing a computer or video game. It usually involves wearing a headset over the eyes and using a controller or remote to interact with the VR content. The content for this study is a guided meditation application. Guided meditation is a relaxation technique used to provide stress relief and reduce tension. A teacher, video, or audio recording is used to help focus on breathing, pleasant scenery, or music.

Intervention 2 will be changes to the procedure room environment. These will include nature imagery and a selection of music. You will be able to choose from a selection of music stations or to pick your favorite type of music to listen to before and during the procedure. Music therapy and nature imagery help provide stress relief and promote relaxation.

There is a 50% chance you will be assigned to one of these interventions. There is also a 50% chance you will be assigned to a control group. Control group participants will receive normal standard of care during their procedure and be asked to answer questions about their experience.

Abbreviated Title: Improving Patient Experience:

**BMBA** 


Version Date: 01/10/2022

Version Number: 1.1

# **Procedures**

124

123

125 While you are in this study, you will have your bone marrow biopsy procedure as part of your 126 normal care. Please note that additional tests and procedures are not expected but may be 127 needed to check on your health condition.

128

129 Name of Procedure: Bone Marrow Biopsy / Aspiration

130

131 Description: After numbing the procedure area with lidocaine, a small fragment of bone will be 132 removed along with a small sample of marrow using a needle. This will be done one time during 133 your visit.

134

135 Name of Evaluation: Vital Signs

136

137 Description: Before your bone marrow biopsy procedure, your heart rate, blood pressure, and 138 respiratory rate will be recorded. Each will be taken once before your procedure.

139 140

**Risks** 

141 142

Taking part in this study involves certain risks. There may be different risks depending on what group you are assigned to. There may also be risks that are not known at this time. If you have any medical issues during this study, call the appropriate number in the contacts section of this form.

145 146 147

143

144

Intervention 1: Virtual reality may cause symptoms associated with motion sickness, including nausea, dizziness, disorientation, and vertigo. Mild eyestrain or headaches may also occur.

148 149 150

Intervention 2: There are no known risks associated with music therapy or décor changes.

151 152

# **Research-Related Injury**

153 154

155

156

157

158

159

160

161

There is a possibility that you could have research-related injury, which is an illness or an injury that is directly caused by the study interventions or a study procedure. If you have a researchrelated injury, we will offer you reasonable and necessary care to treat injuries directly resulting from taking part in this research. Neither Jefferson nor the study will pay for costs associated with treatment of research-related injury or illness. These costs may be billed to your insurance. In addition, you will be responsible for any deductibles and co-payments required under your health plan and for any claims ultimately denied by your health plan. There are no plans for Jefferson to pay you or give you other compensation for the injury. If you think you have been injured as a result of taking part in this research study, tell the research personnel as soon as possible. Please see the contact information in this consent form.

Abbreviated Title: Improving Patient Experience:

**BMBA** 

164 165

## **Disclosure of Financial Interest**

166 167

This study has been funded by the DAISY Foundation's J. Patrick Barnes Grant.

168 169

# **Privacy and Confidentiality: HIPAA Authorization**

170 171

172

Information will be collected about you for this study. The information will be seen by the people involved with this research. Steps will be taken to protect your identity. But the information collected about you can never be 100% secure.

Version Date: 01/10/2022

Version Number: 1.1


173 174 175

HIPAA (Health Insurance Portability and Accountability Act) – This is the law that protects your personal health information.

176 177 178

179

180

To do this study, we need to collect, use, and share your personal health information. This form will explain why your information is being collected, what information will be collected, and who will have access to it. By signing, you are giving us permission to use your information as described in this form.

181 182 183

184

185

186

We are committed to respecting your privacy and to keeping your personal health information confidential. Your personal health information includes the information in your health care records and information that can identify you. For example, personal information may include your name, address, phone number, social security number, and medical information. The personal health information that may be collected, used, and shared for this research includes:

187 188

191

192

193

194

195

196

197

• Information from your medical records

189 190

• Demographic information such as name, gender, birth date, ethnicity, medical history, health care providers, race, and ethnicity

 Physical examinations, procedures, tests, labs, your medical conditions, and medications you use

- Information collected about any research related injury
- Information about mental health, sexually transmitted diseases, HIV, AIDS, drug and alcohol use, genetic test results, and other sensitive information
- Vitals, including heart rate, blood pressure, and respiratory rate
- Questionnaires about your experience

198 199 200

Your personal information will be used by and shared with the following:

201 202

203

- Personnel at Thomas Jefferson University and its affiliates for the purpose of this research
- Institutional Review Boards (ethics committees that review research) including the Jefferson IRB

Abbreviated Title: Improving Patient Experience:

**BMBA** 

• Health insurance providers

• Public health authorities who monitor such things as sexually transmitted diseases, HIV, AIDS, child abuse, as required by law

Version Date: 01/10/2022

Version Number: 1.1


- Groups monitoring the safety of the study such as a data and safety monitoring committee
- Others as required by law

209210211

212

213

214

215

206

207

208

When your personal information is provided to some of the people listed, it may no longer be protected under the HIPAA privacy law. You can see your health care records at any time. However, generally you will not be able to see your study records or the study results until the study is completed. A copy of this signed form, information about this study, and the results of any study test or procedure may be included in your health records which may be seen by your insurance company and your health care providers.

216217218

This authorization does not have an expiration date. Please inform the investigator in writing if you want to end your permission to collect information/samples. Please note that anything already collected will still be used and you may not be able to continue in this study.

220221222

219

The information from this study may be published in scientific journals or presented at scientific meetings, but you will not be personally identified.

223224225

A description of this study will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

227228229

226

Your private information, with the identifiers removed, could be used for future research studies or distributed to other researchers for future research studies without your additional permission.

231232233

230

#### Contacts

234235

If you are having a medical emergency, call 911 or go directly to an emergency room. You should let emergency personnel or providers know that you are taking part in this study.

PI: Anne Delengowski, RN, MSN, AOCN, CCCTM IRB Control #: 21G.1035 Abbreviated Title: Improving Patient Experience:

BMBA

| For Questions About: | Person or Office | Contact Information |
|---|---|---|
| The Study or Research Related | Main Investigator: Anne | (215) 955-7098 |
| Injury | Delengowski | |
| | Investigator: Michelle | (267) 438-6652 |
| | Lasota | |
| If you need to contact someone | Jefferson Center City | 215-503-0203 |
| other than the study personnel | | |
| about a concern or your rights as | Institutional Review Board | 215-503-8966 |
| a research subject | (Ethics Committee) | |
| | | 215-955-4239 |

Version Date: 01/10/2022 Version Number: 1.1


Abbreviated Title: Improving Patient Experience:

BMBA

Version Date: 01/10/2022 Version Number: 1.1 Page **8** of **8** 

| Signatures |
|------------|
|------------|

Patient/Subject: By signing this form, you are agreeing that:

244 245

241 242

- You were given the opportunity to read this form.
- All of the information in this form was discussed with you by an investigator or other

| <ul><li>research personnel to yo</li><li>All your questions have b</li></ul> | n this form was discussed with you by a<br>our satisfaction.<br>Deen answered to your satisfaction.<br>and you voluntarily agree to take part in | - |
|---|---|---|
| Your Name | Your <b>Signature</b> | <br>Date |
| Name of Person Obtaining/<br>Assisting with Consent | Signature of Person Obtaining/ Assisting with Consent | <br>Date |
| | ertifies that the study participant has procedures, risks, benefits and alternative | |
| | Signature of Witness nguage the subject speaks and understone f the subject is blind or cannot physically | _ |
| | THOMAS JEFFERSON U | NIVERSITY |
| | . DDD 07117 D 177 1070 | 2021 |
| | APPROVAL DATE 10/28 | /2021 |
| | APPROVAL DATE 10/28/ Approved until END OF S | |